CLINICAL TRIAL: NCT00267748
Title: A Randomized Phase II Study Of The Efficacy And Safety Of Sunitinib Malate Schedule 4/2 vs. Sunitinib Malate Continuous Dosing As First-Line Therapy For Metastatic Renal Cell Cancer (Renal EFFECT Trial)
Brief Title: Sunitinib Malate Schedule 4/2 vs. Sunitinib Malate Continuous Dosing As First-Line Therapy For Metastatic Renal Cell Cancer (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181065
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-08

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (Experimental)
  Interventions: Drug: Sunitinib Malate Continuous Daily Dosing
- A (Experimental)
  Interventions: Drug: Sunitinib Malate Schedule 4/2

INTERVENTIONS:
Drug: Sunitinib Malate Continuous Daily Dosing — Sunitinib malate starting dose 37.5 mg daily continuous daily regimen.
  Arms: C
Drug: Sunitinib Malate Schedule 4/2 — Sunitinib malate starting dose 50 mg per day for four weeks, followed by a two week off-drug period. This six week cycle is repeated.
  Arms: A

SUMMARY:
This trial has two parts. The purpose of the first part of the trial is to determine the doses of 2 drugs, sunitinib malate and interferon alfa-2b, that can be given safely in combination. This part is currently closed to enrollment.

The purpose of the second part of the trial is to see if sunitinib malate given on a 4/2 schedule (4 weeks on treatment, 2 weeks off treatment cycle) is any better at delaying progression of renal cell cancer than sunitinib malate given on a continuous dosing schedule. The trial will also determine the number of patients whose cancer responds to the treatments, whether life of patients can be extended, what the side effects are of the treatments, how bothersome disease or treatment-related symptoms are to patients, and whether tests can be found that will predict which patients may or may not respond to these treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell carcinoma of clear cell origin or a component of clear cell histology.
* Measurable disease

Exclusion Criteria:

* Prior systemic therapy of any kind for advanced renal cell cancer
* History of brain metastases
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2005-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (117):
- United States (117):
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Baldwin Park, California
  - Pfizer Investigational Site, Bellflower, California
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Fontana, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Panorama City, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Woodland Hills, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Pueblo, Colorado
  - Pfizer Investigational Site, Thorton, Colorado
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Delray Beach, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Jefferson, Indiana
  - Pfizer Investigational Site, Kokomo, Indiana
  - Pfizer Investigational Site, La Porte, Indiana
  - Pfizer Investigational Site, Michigan City, Indiana
  - Pfizer Investigational Site, Plymouth, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Holland, Michigan
  - Pfizer Investigational Site, Niles, Michigan
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Washington, Missouri
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Hackensack, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Farmington, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Amsterdam, New York
  - Pfizer Investigational Site, Brockport, New York
  - Pfizer Investigational Site, Canadaigua, New York
  - Pfizer Investigational Site, Geneva, New York
  - Pfizer Investigational Site, Hudson, New York
  - Pfizer Investigational Site, Latham, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rexford, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Elizabeth City, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Springfield, Oregon
  - Pfizer Investigational Site, Dunmore, Pennsylvania
  - Pfizer Investigational Site, Lemoyne, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Scranton, Pennsylvania
  - Pfizer Investigational Site, Easley, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Seneca, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Round Rock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Hampton, Virginia
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Williamsburg, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Motzer RJ, Hutson TE, Hudes GR, Figlin RA, Martini JF, English PA, Huang X, Valota O, Williams JA. Investigation of novel circulating proteins, germ line single-nucleotide polymorphisms, and molecular tumor markers as potential efficacy biomarkers of first-line sunitinib therapy for advanced renal cell carcinoma. Cancer Chemother Pharmacol. 2014 Oct;74(4):739-50. doi: 10.1007/s00280-014-2539-0. Epub 2014 Aug 7. PMID 25100134
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181065&StudyName=Sunitinib%20Malate%20Schedule%204/2%20vs.%20Sunitinib%20Malate%20Continuous%20Dosing%20As%20First-Line%20Therapy%20For%20Metastatic%20Renal%20Cell%20Cancer%20%28RCC%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib 37.5 mg + Interferon Alpha-2b: Sunitinib 37.5 mg or 50 mg self administered orally once daily in the evening for 4 consecutive weeks followed by 2 weeks off (Schedule 4/2) to comprise a complete 6-weeks cycle. Concomitant Interferon (IFN) alpha-2b self-administered at a dose of 3 million units (MU) or 6 MU or 9MU subcutaneously (s.c.) 3 times weekly on non-consecutive days for up to 1 year (9 cycles) of treatment or early withdrawal.
- Sunitinib 50 mg (Schedule 4/2): Sunitinib 50 mg self administered orally, once daily in the morning for 4 consecutive weeks followed by 2 weeks off treatment to comprise a complete 6-weeks cycle.
- Sunitinib 37.5 mg: Sunitinib 37.5 mg continuous daily dosing (CDD) self administered orally once daily in the morning.
Period: Non-randomized Period
Arm/Group | Sunitinib 37.5 mg + Interferon Alpha-2b | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Started | 25 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 23 | 0 | 0
Not completed — Progressive disease | 10 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Participant not willing to participate | 1 | 0 | 0
Not completed — Other | 3 | 0 | 0
Period: Randomized Period
Arm/Group | Sunitinib 37.5 mg + Interferon Alpha-2b | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Started | 0 | 146 | 146
Treated | 0 | 146 | 143
Completed | 0 | 19 | 14
Not Completed | 0 | 127 | 132
Not completed — Death | 0 | 2 | 3
Not completed — Adverse Event | 0 | 23 | 25
Not completed — Global deterioration of health status | 0 | 6 | 7
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Objective progression or relapse | 0 | 77 | 86
Not completed — Withdrawal by Subject | 0 | 9 | 2
Not completed — Other | 0 | 9 | 6
Not completed — randomized but not treated | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib 37.5 mg + Interferon Alpha-2b | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg | Total
Number analyzed (Participants) | 25 | 146 | 146 | 317
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (7.2) | 60.4 (9.8) | 64.3 (9.7) | 62.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 45 | 57 | 107
  Male | 20 | 101 | 89 | 210

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression (TTP) Assessed Using Memorial Sloan-Kettering Cancer Center (MSKCC) Prognostic Factors Model
Description: MSKCC Prognostic Factor Model assessed as low(0),intermediate(1-2) or high(=>3) based on number of criteria present such as Karnofsky performance status < 80 %, Lactate dehydrogenase > 1.5 * Upper limit of Normal,Hemoglobin < lower limit of normal, serum calcium > 10 mg/dL;Time from first diagnosis of renal cell carcinoma to start of systemic therapy of < 1 year.TTP was time from start of study treatment to first documentation of objective tumor progression or death due to cancer.TTP was calculated as (first event date minus date of first dose of study medication plus 1) divided by 30.44.
Time Frame: From date of randomization until the date of first documented progression or date of death due to any cause, assessed up to a maximum of 2 years
Population: The intent-to-treat (ITT) population included all participants who were randomized into the study regardless of whether they received study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 146 | 146
Months
  Stratified analysis : High Risk (=>3) | 3.1 [0.5 to 10.4] | 4.4 [1.4 to 7.1]
  Stratified analysis : Intermediate Risk (1-2) | 8.0 [5.1 to 11.1] | 7.1 [5.5 to 10.0]
  Stratified analysis : Low Risk (0) | 20.7 [9.9 to 25.2] | 8.4 [7.0 to 21.0]
  Overall unstratified analysis | 9.9 [7.0 to 13.4] | 7.1 [6.8 to 9.7]
Statistical Analysis 1: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For High risk factor, the hazard ratio of TTP was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median TTP was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.860, Log Rank; Hazard Ratio (HR) = 1.089, 95% CI 2-sided [0.423 to 2.803]
Statistical Analysis 2: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For intermediate risk factor, the hazard ratio of TTP was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median TTP was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.583, Log Rank; Hazard Ratio (HR) = 0.902, 95% CI 2-sided [0.623 to 1.306]
Statistical Analysis 3: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For low risk factor, the hazard ratio of TTP was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median TTP was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.075, Log Rank; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.288 to 1.074]
Statistical Analysis 4: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For overall stratified analysis, the hazard ratio of TTP was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median TTP was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.220, Log Rank; Hazard Ratio (HR) = 0.827, 95% CI 2-sided [0.609 to 1.124]
Statistical Analysis 5: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For overall unstratified analysis, the hazard ratio of TTP was estimated using stratified Cox Proportional Hazard model. Two-sided unstratified Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.090, Log Rank; Hazard Ratio (HR) = 0.773, 95% CI 2-sided [0.572 to 1.044]

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with atleast 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized into the study regardless of whether they received study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 146 | 146
Percentage of participants | 32.2 [24.7 to 40.4] | 28.1 [21.0 to 36.1]
Statistical Analysis 1: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; Response rate was estimated for each treatment group, 95% Confidence Interval (CI) on the difference in response rate between the 2 treatments was computed. P-value was calculated from a Pearson chi-square test; Test type: Superiority or Other; p = 0.444, Chi-squared; Mean Difference (Net) = 4.110, 95% CI 2-sided [-6.4 to 14.6]

3. Secondary Outcome: Duration of Response (DR)
Description: Time from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.44. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: DR was calculated for the subgroup of participants from the ITT set, with a confirmed OR.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 47 | 41
Months | 12.5 [1.9 to 23.4] | 8.7 [1.2 to 22.4]

4. Secondary Outcome: Overall Survival (OS) Assessed Using MSKCC Prognostic Factors Model
Description: MSKCC Prognostic Factor Model assessed as low (0), intermediate (1-2) or high (=>3) based upon number of criteria present. Criteria as follows: Karnofsky performance status < 80 %, Lactate dehydrogenase > 1.5 * Upper limit of Normal, Hemoglobin < lower limit of normal for local lab, Corrected serum calcium > 10 mg/dL; Time from first diagnosis of renal cell carcinoma to start of systemic therapy of < 1 year. OS was defined as time from date of start of treatment to date of death due to any cause. OS, in months, was calculated as (event date -start of treatment date + 1)/30.44.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 146 | 146
Months
  High Risk (equal or more than 3) | 3.5 [1.1 to 21.2] | 6.1 [3.6 to 15.1]
  Intermediate Risk (1-2) | 19.3 [14.0 to 24.7] | 21.8 [14.5 to NA] — Higher confidence interval was inevaluable because insufficient participants experienced events
  Low Risk (0) | NA [24.4 to NA] — Insufficient participants experienced events to calculate median | 28.9 [28.9 to NA] — Higher confidence interval was inevaluable because insufficient participants experienced events
Statistical Analysis 1: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For high risk factor, the hazard ratio of OS was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median OS was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.866, Log Rank; Hazard Ratio (HR) = 1.071, 95% CI 2-sided [0.481 to 2.387]
Statistical Analysis 2: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For intermediate risk factor,the hazard ratio of OS was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median OS was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.439, Log Rank; Hazard Ratio (HR) = 1.169, 95% CI 2-sided [0.785 to 1.741]
Statistical Analysis 3: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For low risk factor, the hazard ratio of OS was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median OS was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.614, Log Rank; Hazard Ratio (HR) = 1.238, 95% CI 2-sided [0.538 to 2.851]
Statistical Analysis 4: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; For overall stratified analysis, the hazard ratio of OS was estimated using stratified Cox Proportional Hazard model with the MSKCC prognostic factors (low, intermediate, high), used in the randomization, as a stratum and median OS was estimated using Kaplan-Meier method. Log rank method was used to calculate p value; Test type: Superiority or Other; p = 0.365, Log Rank; Hazard Ratio (HR) = 1.162, 95% CI 2-sided [0.838 to 1.612]

5. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy-General (FACT-G)
Description: FACT-G is core questionnaire of Functional Assessment of Chronic Illness Therapy (FACIT) measurement system to evaluate quality of life (QoL) in cancer population.FACT-G consisted of 27 questions grouped in 4 domains of general Health-Related QoL(HRQoL):Physical Well-being(PWB),Social/Family Well-Being (SWB),Emotional Well-Being (EWB) and Functional Well-Being (FWB);each ranging from 0 (not at all) to 4 (very much) so that FACT-G ranged between 0-108.Since questions could be reversed coded, as appropriate, before calculating FACT-G,0 and 108 could be considered worst and best health states.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 95 | 103
Units on a scale | 78.0 (15.9) | 77.0 (17.1)
Statistical Analysis 1: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; P value was calculated using sample t-test; Test type: Superiority or Other; p = 0.6737, t-test, 2 sided

6. Other Pre Specified Outcome: FACT-Kidney Symptom Index for Disease Related Symptoms (FKSI-DRS)
Description: FKSI-DRS is a subset of FKSI which is a questionnaire for Functional Assessment of Cancer Therapy -Kidney Symptom Index used to assess QoL/participant-reported outcomes for participants diagnosed with renal cell cancer.
  The FKSI contained 15 questions and the FKSI-DRS consisted of 9 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI-DRS ranged between 0-36. Since the questions could be reversed coded, as appropriate, before calculating FKSI-DRS, 0 and 36 could be considered the worst and best health states based on the 9 questions comprising FKSI-DRS.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Number analyzed (Participants) | 95 | 104
Units on scale | 28.3 (5.6) | 27.2 (5.9)
Statistical Analysis 1: Comparison: Sunitinib 50 mg (Schedule 4/2) vs Sunitinib 37.5 mg; P value was calculated using sample t-test; Test type: Superiority or Other; p = 0.1967, t-test, 2 sided

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib 37.5 mg + Interferon Alpha-2b | Sunitinib 50 mg (Schedule 4/2) | Sunitinib 37.5 mg
Serious Adverse Events (participants affected / at risk) | 7/25 | 50/146 | 54/143
Other Adverse Events (participants affected / at risk) | 25/25 | 144/146 | 142/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg + Interferon Alpha-2b (N=25) | Sunitinib 50 mg (Schedule 4/2) (N=146) | Sunitinib 37.5 mg (N=143)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 2
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 6 | 12
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 1 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Disseminated intravascular coagulati (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 4 | 1
Device dislocation (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 3 | 0
Disease progression (General disorders) | 0 | 7 | 11
Fatigue (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 3
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Subacute endocarditis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 5
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Demyelination (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 4
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Microangiopathy (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg + Interferon Alpha-2b (N=25) | Sunitinib 50 mg (Schedule 4/2) (N=146) | Sunitinib 37.5 mg (N=143)
Fatigue (General disorders) | 25 | 94 | 100
Pyrexia (General disorders) | 8 | 23 | 17
Chills (General disorders) | 7 | 14 | 18
Influenza like illness (General disorders) | 6 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 41 | 36
Oedema peripheral (General disorders) | 2 | 29 | 26
Diarrhoea (Gastrointestinal disorders) | 20 | 85 | 98
Nausea (Gastrointestinal disorders) | 14 | 91 | 76
Stomatitis (Gastrointestinal disorders) | 13 | 32 | 33
Dyspepsia (Gastrointestinal disorders) | 10 | 37 | 36
Vomiting (Gastrointestinal disorders) | 8 | 48 | 48
Constipation (Gastrointestinal disorders) | 5 | 40 | 39
Abdominal pain (Gastrointestinal disorders) | 4 | 16 | 15
Oral pain (Gastrointestinal disorders) | 4 | 19 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 19 | 7
Abdominal distension (Gastrointestinal disorders) | 2 | 12 | 2
Glossitis (Gastrointestinal disorders) | 2 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 2 | 10 | 7
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 7 | 8
Dysgeusia (Nervous system disorders) | 7 | 55 | 49
Dizziness (Nervous system disorders) | 6 | 22 | 20
Headache (Nervous system disorders) | 5 | 33 | 23
Paraesthesia (Nervous system disorders) | 5 | 0 | 0
Ageusia (Nervous system disorders) | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 22 | 20
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 46 | 36
Rash (Skin and subcutaneous tissue disorders) | 6 | 36 | 44
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 10 | 10
Yellow skin (Skin and subcutaneous tissue disorders) | 4 | 8 | 7
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 18 | 21
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 14 | 24 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 35 | 28
Leukopenia (Blood and lymphatic system disorders) | 7 | 8 | 5
Anaemia (Blood and lymphatic system disorders) | 5 | 25 | 27
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 29 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 34 | 25
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 29 | 31
Decreased appetite (Metabolism and nutrition disorders) | 11 | 46 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 20 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 14 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 32 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 29 | 24
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Weight decreased (Investigations) | 3 | 20 | 30
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0
Hypertension (Vascular disorders) | 6 | 46 | 42
Accelerated hypertension (Vascular disorders) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 10 | 8
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 19 | 11
Lacrimation increased (Eye disorders) | 0 | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 11 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 11 | 12
Dysphagia (Gastrointestinal disorders) | 0 | 12 | 5
Flatulence (Gastrointestinal disorders) | 0 | 10 | 12
Haemorrhoids (Gastrointestinal disorders) | 0 | 6 | 8
Toothache (Gastrointestinal disorders) | 0 | 8 | 3
Asthenia (General disorders) | 0 | 13 | 16
Chest pain (General disorders) | 0 | 7 | 8
Pain (General disorders) | 0 | 4 | 13
Sinusitis (Infections and infestations) | 0 | 11 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 12 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 8 | 12
Blood creatinine increased (Investigations) | 0 | 11 | 11
Haemoglobin decreased (Investigations) | 0 | 6 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 10 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 13 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 9 | 9
Anxiety (Psychiatric disorders) | 0 | 14 | 11
Depression (Psychiatric disorders) | 0 | 10 | 18
Insomnia (Psychiatric disorders) | 0 | 27 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 8 | 16
Erythema (Skin and subcutaneous tissue disorders) | 0 | 12 | 7
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 9 | 7
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 10 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.